CLINICAL TRIAL: NCT00913185
Title: Acne Free vs. Proactiv for the Treatment of Moderately Severe Acne Vulgaris
Brief Title: Comparison Study of Topical Acne Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedDerm Associates (Industry)
Responsible Party: Principal Investigator, Michelle Pelle, M.D., Principal Investigator, MedDerm Associates
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1021; NCT00419523 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2009-06-04 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Acne Free, Proactiv

SUMMARY:
The purpose of this study is to compare the effectiveness of two over the counter acne products in subjects with moderate severity acne vulgaris. The two products being compared in this study are Acne Free "Severe Acne Line" manufactured by University Medical Products, and Proactiv® manufactured by Guthy-Renker.

DETAILED DESCRIPTION:
You will receive a study drug for the 8 week study. No subject will be given a placebo (an inactive substance) during treatment.The study drugs (over the counter acne medications) have been previously tested and their safe use has been established. However, not all risks or side effects are known. In rare cases of allergy, side effects may be life threatening.The most common side effects of this study drug are:

1. Dry skin
2. Peeling skin
3. Red skin
4. Burning or tingling (temporary)

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or subjects' legal guardians who understand and are willing to sign an Informed Consent Form, an Assent Form if indicated, and a HIPAA Authorization Form.
* Subjects who have received the permission of a parent or guardian to participate in this study or cannot be classified as a minor, under the age of 18 years.
* Male and female subjects between the ages of 13 and 45 years and in generally good health, as determined by a Medical History Form.
* Subjects with moderately-severe acne vulgaris of the face and neck as determined and defined by baseline lesion counts (see Definition: Acne Severity above).
* Subjects who have completed a Medical History Form.
* Subjects who have not used oral acne medications for 1 month prior to start of study, and topical acne medications 1 week prior to start of study.
* Subjects who agree not to use any acne medication during the study except for the test materials given to them.
* Subjects who agree not to use any make-up that contains acne treatment additives, such as benzoyl peroxide, salicylic acid or retinol.
* Subjects who are willing to be photographed and video-recorded during study visits and willing to sign photographic release forms.
* Subjects who exhibit dependability and intelligence in following directions.

Exclusion Criteria:

* Subjects who are pregnant or lactating.
* Subjects with known allergies to cosmetic, toiletry, or acne treatment products.
* Subjects who are sensitive to any of the ingredients in the test articles.
* Subjects who have participated in a facial treatment study within 3 weeks of study initiation.
* Subjects exhibiting acute or chronic dermatological, medical, and/or physical conditions which would preclude application of the test materials and/or influence the outcome of the study.
* Subjects who are unable to sit quietly for 15 minutes to acclimate to ambient temperature and humidity conditions in the laboratory.
* Male subjects who do not have a full beard.
* Subjects who cannot stop usage of oral acne mediation 1 month prior to study start, and topical acne medications 1 week prior to study start.
* Subjects taking routine high dosage anti-inflammatory medications (aspirin, ibuprofen).
* Subjects who must use oral corticosteroids and/or oral immunosuppressive drugs (steroid inhalers or decongestant nose drops and/or eye drops are permitted).
* Any condition for which the Investigator determines that the subject could be placed under undo risk.

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle T Pelle, M.D., Principal Investigator — Medical Director
Locations (1):
- MedDerm Associates, San Diego, California, United States

REFERENCES:
- See also: Related Info — http://medderm.net